CLINICAL TRIAL: NCT05104684
Title: Chest Physical Therapy in Patients Waiting for Allogeneic Hematopoietic Stem Cell
Brief Title: Chest Physical Therapy in Patients Waiting for Allogeneic Hematopoietic Stem Cell Transplantation"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ZIZI MOHAMMED IBRAHIM ALI, Assistant Professor of physical therapy, Department of Physical Therapy for Burn and Plastic Surgery, Faculty of Physical Therapy, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stem cell
Record Dates: First submitted 2021-10-09; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Fifty patients scheduled for HSCT at the bone marrow transplant will randomly be assigned into two groups; one will receive Chest Physical Therapy in addition to routine medical treatment and the control group will receive routine medical treatment only. Outcomes will be a pulmonary function that will be measured by spirometry and respiratory muscle strength measure by Respiratory Pressure Meter. Measurements will be before three weeks before then at the end of treatment immediately before Hematopoietic Stem Cell Transplantation and the last assessment at three weeks after hematopoietic Stem Cell Transplantation for all measured variables..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A:Chest Physical Therapy (Experimental): Patients in group A will receive CPT program daily for three weeks before HSCT (hospital stay for allogeneic-HCT). The program consists of postural drainage, diaphragmatic breathing exercises, coughing, huffing, percussion, shaking, and exercise training using an incentive spirometer in addition to routine medical treatment. The total duration of each CPT session ranged from 45-60 minutes according to patient tolerance. The choice of airway clearance method that will be applied depends on two factors; patient preference and the individual response of the patient to treatment.
  Interventions: Other: chest physical therapy; Other: routine medical treatment
- Control group (B):Routine medical treatment (Active Comparator): patients in group B will receive routine medical treatment
  Interventions: Other: routine medical treatment

INTERVENTIONS:
Other: chest physical therapy — The program will consist of postural drainage, diaphragmatic breathing exercises, coughing, huffing, percussion, shaking, and exercise training using an incentive spirometer in addition to routine medical treatment
  Other Names: chest p.t
  Arms: group A:Chest Physical Therapy
Other: routine medical treatment — medical treatment

SUMMARY:
evaluate the efficacy of Chest Physical Therapy (CPT) performed during the pre-transplant period on spirometric values as well as Respiratory Muscle Strength (RMS) in patients waiting for Allogeneic Hematopoietic Stem Cell Transplantation

DETAILED DESCRIPTION:
patients scheduled for HSCT at the bone marrow transplant will randomly be assigned into two groups; one will receive Chest Physical Therapy in addition to routine medical treatment and the control group will receive routine medical treatment only. Outcomes will be a pulmonary function that will be measured by spirometry and respiratory muscle strength measure by Respiratory Pressure Meter. Measurements will be before three weeks before then at the end of treatment immediately before Hematopoietic Stem Cell Transplantation and the last assessment at three weeks after hematopoietic Stem Cell Transplantation for all measured variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively admitted to HSCT unit, completed the induction therapy and awaiting for allogeneic HSCT Study. Candidates' ages from 40-55 years old, both males and females will be included, Non-smokers patients, Non-alcoholics patients, patients medically cleared to exercise that decided by the transplant physician; patients able to understand training instructions and follow the study protocol

Exclusion Criteria:

* fever
* smokers

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Spirometry measures1 | Change from Baseline (three weeks before HSCT) , the end of treatment immediately before HSCT(T1) to three weeks after HSCT(T2) for all measured variables.
  The forced expiratory volume in one second (FEV1), FEV1 is the volume of air exhaled in the first second of the FVC maneuver
Spirometry measures2 | Change from Baseline (three weeks before HSCT) , the end of treatment immediately before HSCT(T1) to three weeks after HSCT(T2) for all measured variables.
  the forced vital capacity (FVC)To measure FVC, the patient inhales maximally, then exhales as rapidly and as completely as possible.
Spirometry measures3 | Change from Baseline (three weeks before HSCT) , the end of treatment immediately before HSCT(T1) to three weeks after HSCT(T2) for all measured variables.
  the relation between FEV1 and FVC

SECONDARY OUTCOMES:
Respiratory muscle strength (RMS) | A baseline assessment will be done three weeks before HSCT (T0) then at the end of treatment immediately before HSCT(T1) and the last assessment at three weeks after HSCT(T2) for all measured varibles.
  Maximal inspiratory pressure (MIP or PImax) and maximal expiratory pressure (MEP or PEmax) will be measured to assess respiratory muscle strength (RMS) using MicroMedical MicroRPM 01 (Respiratory Pressure Meter) according to ATS/ERS guidelines

CONTACTS AND LOCATIONS:
Overall Officials: INTSAR S WAKED, PHD, Principal Investigator — Cairo University
Locations (1):
- Zizi Mohammed Ibrahim Ali, Giza, Nnjkjk, Egypt

IPD SHARING:
Plan to Share IPD: Undecided